CLINICAL TRIAL: NCT03502200
Title: Switching to a Vaping Device: Evaluating Risk Reduction Among Quitline Treatment Failure
Brief Title: Switching to a Vaping Device: Evaluating Risk Reduction Among Quitline Treatment Failures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Theodore Wagener, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-19133; U01DA045537 (NIH)
Record Dates: First submitted 2018-02-28; First posted 2018-04-18 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-06

CONDITIONS: Smoking, Cigarette
Keywords: e-cigarettes; harm reduction; smoking behavior
MeSH Terms: conditions — Cigarette Smoking; Vaping; Harm Reduction; Smoking | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two conditions randomly.
Masking Description: This study is a comparative randomized study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- E-cigarette (Experimental): 5% nicotine JUUL e-cigarette (Tobacco or Menthol flavor). Will also receive counseling.
  Interventions: Device: JUUL
- Treatment As Usual (Active Comparator): Nicotine Replacement Therapy consisting of nicotine patches and lozenge along with standard assessments. Will also receive counseling.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Device: JUUL — Participants randomized to the JUUL group will receive either tobacco or menthol flavored JUUL with 5% nicotine. Will also receive counseling.
  Arms: E-cigarette
Other: Treatment As Usual — Nicotine Replacement Therapy consisting of nicotine patches and lozenge along with standard quitline counseling.
  Arms: Treatment As Usual

SUMMARY:
The overall aim of the study is to evaluate the provision of e-cigarette (EC) versus NRT on smoking behavior, product use patterns and continued use, and iCO, a biomarker of toxicant exposure, among a sample of recent QL treatment failures. We will randomly assign N=372 smokers (targeted accrual) to EC (n=186) or QL treatment as usual with combination nicotine replacement therapy (NRT; n=186). All participants will receive three calls from QL coaches and EC and NRT will be provided at no cost for 8 weeks. The final follow-up will occur 12-weeks post baseline.

DETAILED DESCRIPTION:
There remains a lack of prospective and controlled research on the behavioral, toxicological, and physiological effects of electronic cigarettes (ECs) to help the public health community come to a clear and accurate consensus on their risk-benefit. In order to successfully execute the proposed study, the investigators plan to recruit and enroll recent smoking cessation treatment failures from a state QL, which predominately serves priority populations (e.g., low socioeconomic status, high levels of mental health conditions). The proposed study will randomly assign smokers who were recent QL treatment failures to a) EC (JUUL 5%) or b) QL treatment as usual with combination nicotine replacement therapy control (NRT).

ELIGIBILITY:
Inclusion Criteria:

* smoke ≥5 cigarettes per day for the past year
* read, write, and speak in English
* report at least minimal interest in switching to an alternative product (> "not at all" on a Likert scale)
* participation in the Oklahoma Tobacco Helpline or South Carolina Tobacco Helpline within the last 4-7 months.

Exclusion Criteria:

* <21 years old
* report NRT use or making a quit attempt within the last 7 days
* current daily use of an e-cigarette over last month.
* unstable or significant medical condition such as respiratory, kidney, or liver disease
* unstable or significant psychiatric conditions (past and stable conditions will be allowed)
* history of cardiac event or distress within the past 6 months
* currently pregnant, planning to become pregnant, or breastfeeding.
* currently enrolled in a contradictory study.
* cohabitates with a currently enrolled participant in the REACH study
* reaction to using patch medication or adhesive tape
* known allergy to propylene glycol or vegetable glycerin

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore L Wagener, PhD, Principal Investigator — Ohio State Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
De-identified and aggregated data will be shared through poster presentations and published manuscripts.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | E-cigarette | Treatment As Usual
Started | 175 | 175
Completed | 132 | 127
Not Completed | 43 | 48
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 36 | 38
Not completed — Study Team Decision | 1 | 1
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E-cigarette | Treatment As Usual | Total
Number analyzed (Participants) | 175 | 175 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was not collected for 4 participants
  years
    number analyzed (Participants) | 173 | 173 | 346
    (all) | 55.26 (12.66) | 54.19 (12.47) | 54.72 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex was not collected for 4 participants
  Participants
    number analyzed (Participants) | 173 | 173 | 346
    Female | 107 | 105 | 212
    Male | 66 | 68 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 170 | 171 | 341
  Unknown or Not Reported | 3 | 2 | 5
Cigarettes Smoked per Day [Mean (Standard Deviation); unit: cigarettes per day] — Population: 5 Participants were missing data on cigarettes per day smoked at baseline
  cigarettes per day
    number analyzed (Participants) | 172 | 173 | 345
    (all) | 16.78 (8.16) | 17.41 (8.21) | 17.10 (8.18)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Self-Reported 7-day Point Prevalence Abstinence From Cigarettes
Description: Self-Reported 7-day Point Prevalence Abstinence from Cigarettes to assess complete product switching/substitution.
Time Frame: Daily for 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 175 | 175
Participants | 41 | 33

2. Primary Outcome: Proportion of Participants With iCO (Portable Carbon Monoxide Monitor) Verified Abstinence
Description: Intent to treat biochemically verified abstinence rates - participants reporting both 7-day point prevalence abstinence and an iCO reading less than or equal to 8. A portable exhaled carbon monoxide detector confirms daily smoking status. Used to evaluate changes iCO, a biomarker of tobacco constituent exposure and other health effects.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 175 | 175
Participants | 22 | 17

3. Secondary Outcome: Sociodemographic Questionnaire - Age
Description: Assess participant age from the sociodemographic questionnaire
Time Frame: Baseline
Population: Participants who completed the baseline survey; age was not collected for 4 participants
Measure: Mean (Standard Deviation); unit: years
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 173 | 173
years | 55.26 (12.66) | 54.19 (12.47)

4. Secondary Outcome: Sociodemographic Questionnaire - Sex
Description: Assess participant sex from the sociodemographic questionnaire
Time Frame: Baseline
Population: Participants who completed the baseline survey; sex was not collected for 4 participants
Measure: Count of Participants; unit: Participants
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 173 | 173
Participants
  Male | 66 | 68
  Female | 107 | 105

5. Secondary Outcome: Sociodemographic Questionnaire - Marital Status
Description: Assess participant marital status from the sociodemographic questionnaire
Time Frame: Baseline
Population: Participants who completed the baseline survey; marital status was not collected for 4 participants
Measure: Count of Participants; unit: Participants
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 173 | 173
Participants
  Married | 55 | 56
  Divorced/Separated | 50 | 46
  Widowed | 23 | 23
  Not married, but living with romantic partner | 16 | 18
  Romantic partner (not living with) | 5 | 5
  Never married and not in current romantic relationship | 24 | 25

6. Secondary Outcome: Sociodemographic Questionnaire - Ethnicity
Description: Assess participant ethnicity from the sociodemographic questionnaire
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 175 | 175
Participants
  Hispanic or Latino | 2 | 2
  Not Hispanic or Latino | 170 | 171
  Unknown or Not Reported | 3 | 2

7. Secondary Outcome: Sociodemographic Questionnaire - Employment Status
Description: Assess participant employment status from the sociodemographic questionnaire
Time Frame: Baseline
Population: Participants who completed the baseline survey; employment data was not collected for 4 participants; 2 additional participants refused to answer the employment items
Measure: Count of Participants; unit: Participants
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 172 | 172
Participants
  Employed by others part-time for wages | 8 | 12
  Employed by other full-time for wages | 26 | 32
  Self-employed | 11 | 13
  Out of work | 17 | 21
  Homemaker | 11 | 3
  Retired | 30 | 31
  Unable to work/Disabled | 69 | 60

8. Secondary Outcome: Sociodemographic Questionnaire - Socioeconomic Status
Description: Assess participant socioeconomic status via yearly household income
Time Frame: Baseline
Population: Participants who completed the baseline survey; household income was not collected for 4 participants; 7 additional participants refused to answer the income item
Measure: Count of Participants; unit: Participants
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 170 | 169
Participants
  <$35,000 | 136 | 136
  ≥$35,000 | 34 | 33

9. Secondary Outcome: Cigarette/EC Dependency Scale
Description: Assess e-cigarette and cigarette dependence.
  Scores range from 5 to 25 with higher scores indicating a greater level of dependence.
Time Frame: 12 weeks
Population: Participants who completed their 12 week visit and provided responses to each item on the cigarette/e-cigarette dependency scale questionnaire.
  Participants in the treatment as usual arm were not assessed with the e-cigarette dependence scale as it is only applicable to the e-cigarette arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 121 | 124
units on a scale
  Cigarette Dependence Scale | 14.42 (4.51) | 14.11 (4.60)
  e-Cigarette Dependence Scale: number analyzed (Participants) | 112 | 0
  e-Cigarette Dependence Scale | 12.63 (4.99) |

10. Secondary Outcome: Drug Effects/Liking Questionnaire
Description: Assess the desire and liking of products, positive and negative effects (i.e., side effects), and perceived strength and effectiveness
  Scores range from 1 to 5 with higher scores indicating greater strength (effect from smoking cigarettes/vaping e-cigarettes) or liking (liking of effect from smoking cigarettes/vaping e-cigarettes)
Time Frame: 12 weeks
Population: Participants who responded to the drug effects liking questionnaire within 1 week of their week 12 visit.
  Participants in the treatment as usual arm were not assessed with the e-cigarette drug effects and liking questionnaires as they are only applicable to the e-cigarette arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 74 | 66
score on a scale
  Effect from smoking cigarettes | 2.81 (1.32) | 3.20 (1.30)
  Liking of effect after smoking cigarettes | 3.16 (1.17) | 2.97 (1.23)
  Effect from vaping e-cigarette: number analyzed (Participants) | 74 | 0
  Effect from vaping e-cigarette | 2.80 (1.10) |
  Liking of effect from vaping e-cigarette: number analyzed (Participants) | 74 | 0
  Liking of effect from vaping e-cigarette | 3.39 (1.07) |

11. Secondary Outcome: Cigarette Purchase Task - Breakpoint
Description: Asks participants how much they would be willing to pay (ranging from 0¢ to $1,120) for a puff of their own brand cigarette. Specifically they will be asked, "How much would you be willing to pay for a puff of your usual cigarette brand?".
Time Frame: Week 1 (Baseline)
Population: Participants who completed the cigarette purchase task at baseline.
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 170 | 167
Dollars | 2.62 (11.16) | 5.96 (27.42)

12. Secondary Outcome: Tiffany-Drobes Questionnaire of Smoking Urges: Brief Form (QSU)
Description: Smoking and vaping urges/craving will be measured using the Tiffany-Drobes Questionnaire of Smoking Urges: Brief Form with a modified version (replacing the word "cigarette" with "e-cigarette") for EC users. This is a 10-item measure where participants rate smoking/vaping-related items on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Similar to previous studies, we will collapse the items into two previously identified factors (Factor 1: strong desire and intention to smoke/vape; Factor 2: anticipation of relief from withdrawal symptoms). Scores are calculated by summing the items and range from 5 to 35 for each of the factors with higher scores indicating greater craving to smoke/vape.
Time Frame: 12 Weeks
Population: Participants who completed their 12 week visit. Participants in the treatment as usual arm were not assessed with the e-cigarette QSU questionnaire as it is only applicable to the e-cigarette arm.
  Participants in the e-cigarette arm were not assessed with the NRT QSU questionnaire as it is only applicable to the treatment as usual arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 128 | 125
score on a scale
  QSU Desire (cigarette) | 12.97 (9.72) | 13.66 (10.38)
  QSU Relief (cigarette) | 10.13 (7.98) | 10.22 (7.37)
  QSU Desire (e-cigarette): number analyzed (Participants) | 119 | 0
  QSU Desire (e-cigarette) | 16.76 (10.71) |
  QSU Relief (e-cigarette): number analyzed (Participants) | 118 | 0
  QSU Relief (e-cigarette) | 11.82 (8.26) |
  QSU Desire (NRT): number analyzed (Participants) | 0 | 115
  QSU Desire (NRT) |  | 10.56 (8.41)
  QSU Relief (NRT): number analyzed (Participants) | 0 | 114
  QSU Relief (NRT) |  | 8.69 (6.84)

13. Secondary Outcome: Minnesota Nicotine Withdrawal Scale
Description: Asses Nicotine withdrawal and smoking craving, anger/irritability, anxiety, depressed mood, restlessness/difficulty concentrating, increased appetite, sleep problems, and somatic symptoms (nausea, constipation, sore throat, dizziness, coughing).
  Scores range from 0 to 4 with higher scores indicating greater levels of withdrawal (MNWS) or more craving to smoke (MNWS Craving).
Time Frame: 12 Weeks
Population: Participants who completed their 12 week visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 128 | 126
score on a scale
  MNWS | 1.24 (1.01) | 1.38 (1.07)
  MNWS Craving | 1.98 (1.54) | 2.22 (1.47)

14. Secondary Outcome: Change in Motivation Rulers (Scale) From Baseline to Week 12
Description: Assess for changes in motivation from baseline to week 12 among participants who continue to smoke. Rulers including importance, confidence, and readiness to quit smoking (3-items total, with a scale ranging from 0 "not at all important/confident/ready" to 10 "extremely important/confident/ready").
  Medians reported are change from baseline [week 12 score - baseline score] where negative values indicate a decrease in motivation over time and positive values indicate an increase in motivation over time.
Time Frame: 12 Weeks
Population: Participants who continued to smoke cigarettes at their week 12 visit and provided responses to both the baseline and 12 week motivation ruler questionnaire.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 83 | 88
score on a scale
  Importance | 0 [-1 to 1] | 0 [-2 to 0]
  Readiness: number analyzed (Participants) | 82 | 87
  Readiness | -0.5 [-2 to 0] | 0 [-3 to 0]
  Confidence | 0 [-2 to 2] | 0 [-2.5 to 2]

15. Other Pre Specified Outcome: Tobacco Use History Questionnaire - Years of Smoking
Description: Assess years of smoking from the tobacco use history questionnaire
Time Frame: Week 1 (baseline)
Population: Participants who completed the tobacco use history questionnaire at baseline
Measure: Mean (Standard Deviation); unit: years
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 171 | 172
years | 34.15 (12.99) | 31.59 (14.45)

16. Other Pre Specified Outcome: Tobacco Use History Questionnaire - Cigarettes Per Day
Description: Assess average number of cigarettes per day with the tobacco use history questionnaire
Time Frame: Week 1 (baseline)
Population: Participants who completed the tobacco use history questionnaire at baseline
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 172 | 173
cigarettes per day | 16.78 (8.16) | 17.41 (8.21)

17. Other Pre Specified Outcome: Tobacco Use History Questionnaire - 24-hour Quit Attempts
Description: Assess number of previous 24-hour quit attempts with the tobacco use history questionnaire
Time Frame: Week 1 (baseline)
Population: Participants who completed the tobacco use history questionnaire at baseline
Measure: Mean (Standard Deviation); unit: quit attempts
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 167 | 170
quit attempts | 0.93 (2.39) | 0.82 (1.71)

18. Other Pre Specified Outcome: Tobacco Use History Questionnaire - Number of Smokers in the Household
Description: Assess number of smokers in the household with the tobacco use history questionnaire
Time Frame: Week 1 (baseline)
Population: Participants who completed the tobacco use history questionnaire at baseline
Measure: Mean (Standard Deviation); unit: people
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 173 | 173
people | 1.59 (0.84) | 1.53 (0.83)

19. Other Pre Specified Outcome: Tobacco Use History Questionnaire - Cigarette Expectance Effects
Description: Assess cigarette expectance effects with the tobacco use history questionnaire
Time Frame: Week 1 (baseline)
Population: Participants who completed the baseline survey
Measure: Count of Participants; unit: Participants
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 173 | 173
Participants
  When I'm angry, a cigarette can help calm me down.: Disagree | 12 | 19
  When I'm angry, a cigarette can help calm me down.: Disagree a little | 9 | 1
  When I'm angry, a cigarette can help calm me down.: Agree a little | 23 | 24
  When I'm angry, a cigarette can help calm me down.: Agree | 129 | 129
  When I'm angry, a cigarette can help calm me down.: Refuse to answer / Don't know | 0 | 0
  Cigarettes are good for dealing with boredom: Disagree | 26 | 27
  Cigarettes are good for dealing with boredom: Disagree a little | 23 | 12
  Cigarettes are good for dealing with boredom: Agree a little | 28 | 33
  Cigarettes are good for dealing with boredom: Agree | 95 | 101
  Cigarettes are good for dealing with boredom: Refuse to answer / Don't know | 1 | 0
  Smoking keeps my weight down: Disagree | 103 | 100
  Smoking keeps my weight down: Disagree a little | 12 | 10
  Smoking keeps my weight down: Agree a little | 22 | 23
  Smoking keeps my weight down: Agree | 33 | 37
  Smoking keeps my weight down: Refuse to answer / Don't know | 3 | 3
  When I'm upset with someone, a cigarette helps me cope: Disagree | 18 | 16
  When I'm upset with someone, a cigarette helps me cope: Disagree a little | 5 | 8
  When I'm upset with someone, a cigarette helps me cope: Agree a little | 26 | 17
  When I'm upset with someone, a cigarette helps me cope: Agree | 124 | 132
  When I'm upset with someone, a cigarette helps me cope: Refuse to answer / Don't know | 0 | 0
  If I have nothing to do, a smoke can help kill time: Disagree | 25 | 28
  If I have nothing to do, a smoke can help kill time: Disagree a little | 14 | 10
  If I have nothing to do, a smoke can help kill time: Agree a little | 28 | 28
  If I have nothing to do, a smoke can help kill time: Agree | 106 | 107
  If I have nothing to do, a smoke can help kill time: Refuse to answer / Don't know | 0 | 0
  When I'm feeling down, a cigarette can really make me feel good: Disagree | 49 | 48
  When I'm feeling down, a cigarette can really make me feel good: Disagree a little | 18 | 23
  When I'm feeling down, a cigarette can really make me feel good: Agree a little | 45 | 36
  When I'm feeling down, a cigarette can really make me feel good: Agree | 61 | 66
  When I'm feeling down, a cigarette can really make me feel good: Refuse to answer / Don't know | 0 | 0
  Cigarettes keep me from eating more than I should: Disagree | 92 | 85
  Cigarettes keep me from eating more than I should: Disagree a little | 15 | 15
  Cigarettes keep me from eating more than I should: Agree a little | 28 | 23
  Cigarettes keep me from eating more than I should: Agree | 36 | 47
  Cigarettes keep me from eating more than I should: Refuse to answer / Don't know | 2 | 3
  When I'm alone, a cigarette can help me pass the time: Disagree | 31 | 42
  When I'm alone, a cigarette can help me pass the time: Disagree a little | 15 | 12
  When I'm alone, a cigarette can help me pass the time: Agree a little | 30 | 23
  When I'm alone, a cigarette can help me pass the time: Agree | 96 | 95
  When I'm alone, a cigarette can help me pass the time: Refuse to answer / Don't know | 1 | 1
  Smoking cigarettes calms me down when I feel nervous: Disagree | 13 | 15
  Smoking cigarettes calms me down when I feel nervous: Disagree a little | 3 | 10
  Smoking cigarettes calms me down when I feel nervous: Agree a little | 32 | 21
  Smoking cigarettes calms me down when I feel nervous: Agree | 125 | 126
  Smoking cigarettes calms me down when I feel nervous: Refuse to answer / Don't know | 0 | 1
  Smoking helps me control my weight: Disagree | 110 | 109
  Smoking helps me control my weight: Disagree a little | 17 | 15
  Smoking helps me control my weight: Agree a little | 16 | 17
  Smoking helps me control my weight: Agree | 26 | 29
  Smoking helps me control my weight: Refuse to answer / Don't know | 4 | 3

20. Other Pre Specified Outcome: Tobacco Use History Questionnaire
Description: Assess frequency of use all of nicotine/tobacco products including cigars, cigarillos, little cigars, smokeless tobacco, EC, and hookah.
Time Frame: Week 1 (Baseline)
Population: Participants who completed the baseline survey
Measure: Count of Participants; unit: Participants
Arm/Group | E-cigarette | Treatment As Usual
Number analyzed (Participants) | 173 | 173
Participants
  e-cigarette: Daily or almost daily | 2 | 2
  e-cigarette: Less than daily, but at least once a week | 6 | 2
  e-cigarette: Less than weekly, but at least once a month | 13 | 7
  e-cigarette: Less than monthly | 12 | 13
  e-cigarette: Not at all | 139 | 149
  e-cigarette: Refuse to answer/Don't know | 1 | 0
  Cigar: Daily or almost daily | 1 | 0
  Cigar: Less than daily, but at least once a week | 1 | 1
  Cigar: Less than weekly, but at least once a month | 2 | 1
  Cigar: Less than monthly | 11 | 5
  Cigar: Not at all | 158 | 166
  Cigar: Refuse to answer/Don't know | 0 | 0
  Cigarillo: Daily or almost daily | 2 | 3
  Cigarillo: Less than daily, but at least once a week | 5 | 5
  Cigarillo: Less than weekly, but at least once a month | 7 | 2
  Cigarillo: Less than monthly | 8 | 9
  Cigarillo: Not at all | 151 | 153
  Cigarillo: Refuse to answer/Don't know | 0 | 1
  Little Cigar: Daily or almost daily | 2 | 1
  Little Cigar: Less than daily, but at least once a week | 1 | 1
  Little Cigar: Less than weekly, but at least once a month | 0 | 0
  Little Cigar: Less than monthly | 5 | 3
  Little Cigar: Not at all | 165 | 168
  Little Cigar: Refuse to answer/Don't know | 0 | 0
  Smokeless Tobacco: Daily or almost daily | 4 | 1
  Smokeless Tobacco: Less than daily, but at least once a week | 1 | 4
  Smokeless Tobacco: Less than weekly, but at least once a month | 0 | 3
  Smokeless Tobacco: Less than monthly | 2 | 1
  Smokeless Tobacco: Not at all | 166 | 164
  Smokeless Tobacco: Refuse to answer/Don't know | 0 | 0
  Hookah: Daily or almost daily | 0 | 0
  Hookah: Less than daily, but at least once a week | 0 | 1
  Hookah: Less than weekly, but at least once a month | 0 | 2
  Hookah: Less than monthly | 0 | 2
  Hookah: Not at all | 172 | 168
  Hookah: Refuse to answer/Don't know | 1 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | E-cigarette | Treatment As Usual
All-Cause Mortality (participants affected / at risk) | 0/175 | 2/175
Serious Adverse Events (participants affected / at risk) | 18/175 | 10/175
Other Adverse Events (participants affected / at risk) | 93/175 | 87/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E-cigarette (N=175) | Treatment As Usual (N=175)
Breast Cancer (Reproductive system and breast disorders) | 2 | 0
Breathing Difficulties (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Broken Back (Musculoskeletal and connective tissue disorders) | 0 | 1
Carotid Endarterectomy Surgery (Surgical and medical procedures) | 0 | 1
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest Pain (Cardiac disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Cuff Repair Surgery (Blood and lymphatic system disorders) | 1 | 0
Dental Problems (Surgical and medical procedures) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Essential Tremor Worsening (Nervous system disorders) | 1 | 0
Exploratory Larynx Surgery (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gallbladder Problems (Hepatobiliary disorders) | 1 | 0
Gastrointestinal Problems (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Heart Condition (Cardiac disorders) | 1 | 0
Heart Palpitations (Cardiac disorders) | 1 | 1
Hernia (Surgical and medical procedures) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Needed Medication Adjustment for Bipolar Schizoaffective Disorder (Psychiatric disorders) | 1 | 0
Pancreatic Pain (Gastrointestinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Suicidal Thoughts (Psychiatric disorders) | 1 | 1
Ulcer (Gastrointestinal disorders) | 0 | 2
Wound Abscess (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E-cigarette (N=175) | Treatment As Usual (N=175)
Allergies (Immune system disorders) | 2 | 21
Breathing Difficulties (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 52 | 17
Dizziness (Nervous system disorders) | 10 | 23
Headache (Blood and lymphatic system disorders) | 20 | 23
Mouth or Tongue Sores or Inflammation (Gastrointestinal disorders) | 10 | 14
Sleeplessness (Psychiatric disorders) | 9 | 21
Sore or Dry Mouth and Throat (Gastrointestinal disorders) | 46 | 36
Sleepiness (Nervous system disorders) | 5 | 11
Sleeplessness (Nervous system disorders) | 5 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT03502200/Prot_SAP_ICF_000.pdf